CLINICAL TRIAL: NCT06475261
Title: Tissue Oximetry's Measurement in Cytoreductive Surgery With Hyperthermic Intraperitoneal Chemotherapy: Prospective Observational Study With Device
Brief Title: Tissue Oximetry's Measurement in Cytoreductive Surgery With Hyperthermic Intraperitoneal Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6702
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Oxygen Deficiency; Acute Kidney Injury; Ovarian Carcinoma
Keywords: Tissue Oximetry; Hyperthermic Intraperitoneal Chemotherapy; Acute Kidney Injury; Hemodynamics parameters
MeSH Terms: conditions — Hypoxia; Acute Kidney Injury; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tissue Oximetry with ForeSight — Evaluation of a correlation between average intraoperative muscle tissue oximetry and postoperative renal damage in patients undergoing cytoreductive surgery with HIPEC for ovarian cancer
  Other Names: Hemodynamics parameters with Hemosphere

SUMMARY:
Tissue oximetry obtained from peripheral muscle measures the state of tissue oxygenation of various organs and, as already widely described in the literature, can be used to measure the state of kidney's tissue oxygenation. However, there is no evidence in the existing scientific literature on the use of muscle tissue oximetry in patients undergoing cytoreductive surgery for ovarian cancer with hyperthermic intraperitoneal chemotherapy.

The primary objective of our study is to evaluate whether there is a correlation between average intraoperative muscle tissue oximetry below 65% (a value which is considered critical in the literature for the resulting cellular damage) and postoperative renal damage in patients undergoing cytoreductive surgery with hyperthermic intraperitoneal chemotherapy for ovarian cancer.

DETAILED DESCRIPTION:
Tissue oximetry obtained from peripheral muscle can be used to measure the state of kidney's tissue oxygenation.

50 Adult female patients ASA 1-2 undergoing cytoreductive surgery with laparoscopic or laparotomy technique (for ovarian cancer) associated with hyperthermic intraperitoneal chemotherapy will be enrolled.

The primary objective of our study is to evaluate whether there is a correlation between average intraoperative muscle tissue oximetry below 65% (a value which is considered critical in the literature for the resulting cellular damage) and postoperative renal damage (according to the AKIN and KIDGO classification) in patients undergoing cytoreductive surgery with hyperthermic intraperitoneal chemotherapy for ovarian cancer.

Secondary objectives are:

* describe the variation in muscle tissue oximetry and hemodynamic parameters (systolic, mean, diastolic blood pressure) during cytoreductive surgery with hyperthermic intraperitoneal chemotherapy .
* describe the variation in renal function values (blood urea nitrogen, creatinine) and serum electrolytes (sodium, potassium, chloremia, calcemia) in the post-operative period (from the first to the seventh postoperative day).

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiologists (ASA) Classification 1-2
* Cytoreductive surgery for ovarian cancer with laparoscopic or laparotomic technique with Hypertermic Intraperitoneal Chemotherapy.

Exclusion Criteria:

* Age < 18 years
* ASA > or = 3
* Cytoreductive surgery without hyperthermic intraperitoneal chemotherapy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients ASA 1-2 undergoing cytoreductive surgery with laparoscopic or laparotomy technique (for ovarian cancer) associated with hyperthermic intraperitoneal chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-27 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between intraoperative tissue oximetry and postoperative acute renal injury. | Tissue oximetry is defined as TWA (time-weighted average) value resulted by values recorded intraoperatively every 20 minutes.
  An intraoperative mean tissue oximetry value of 65% or less is considered to predict cellular damage. Postoperative renal injury is classified according to AKIN and KIDGO criteria.

SECONDARY OUTCOMES:
Tissue oximetry | TWA value resulted by intraoperative values recorded every 20 minutes during surgery.
  Describing intraoperative variation of tissue oximetry expressed in percent.
Tissue oximetry during hyperthermic intraperitoneal chemotherapy | TWA value resulted by intraoperative values recorded every 20 minutes during hyperthermic intraperitoneal chemotherapy .
  Describing variation of tissue oximetry during hyperthermic intraperitoneal chemotherapy, expressed in percent.
Emodinamic parameters (systolic, mean and diastolic pressures) | Intraoperatively, a mean value resulted by values recorded every 20 minutes during surgery.
  Describing mean values of intraoperative arterial pressure (systolic, mean and diastolic pressures), expressed in mmHg
Emodinamic parameters (systolic, mean and diastolic pressures) during hyperthermic intraperitoneal chemotherapy | A mean value resulted by values recorded every 20 minutes during hyperthermic intraperitoneal chemotherapy
  Describing mean values of arterial pressure (systolic, mean and diastolic pressures), expressed in mmHg, during hyperthermic intraperitoneal chemotherapy
Serum Creatinine level | From 1st to 7th postoperative days
  Mean value of creatinine, daily assessed for the first 7 postoperative days, expressed in mg/dL
Serum Blood urea nitrogen level | From 1st to 7th postoperative day
  Mean value of Serum blood urea nitrogen, daily assessed for the first 7 postoperative days, expressed in mg/dL
Serum sodium level | From 1st to 7th postoperative day
  Mean values of Serum sodium, daily assessed for the first 7 postoperative days, expressed in mmol/L
Serum Potassium level | From 1st to 7th postoperative day
  Mean values of Serum potassium, daily assessed for the first 7 postoperative days, expressed in mmol/L
Serum Chloride level | From 1st to 7th postoperative day
  Mean values of Serum chloride, daily assessed for the first 7 postoperative days, expressed in mmol/L
Serum Calcium level | From 1st to 7th postoperative day
  Mean values of Serum calcium, daily assessed for the first 7 postoperative days, expressed in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Catarci, MD, Principal Investigator — FPG IRCCS
Locations (1):
- Policlinico "A. Gemelli" IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No